CLINICAL TRIAL: NCT05977309
Title: The Effect of Therapy Ozone Topical on The Healing Diabetic Foot Ulcer: A Triple-Blind Randomized Clinical Trial
Brief Title: Effect of Topical Ozone on The Healing Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asmat Burhan (Other)
Responsible Party: Sponsor-Investigator, Asmat Burhan, Chief Researcher in Nursing, Faculty of Health Sciences, Universitas Harapan Bangsa, Universitas Harapan Bangsa
Organization: Universitas Harapan Bangsa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHarapanBangsa
Record Dates: First submitted 2023-07-12; First posted 2023-08-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Wound Heal; Diabetic Foot Ulcer; Ozone
Keywords: ozone; wound healing; diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: In five wound care clinics on Java Island, Indonesia, 430 men and women with diabetic foot ulcer lesions participated in this randomised, triple-blind clinical trial. Inclusion criteria included women and men receiving treatment for diabetic foot ulcers, the Wagner scale, current blood sugar between 120 and 180 mg/dl, Hb1ac between 4.5 and 7%, lesion length greater than 5 cm, and infection. Exclusion criteria in this investigation, such as immunodeficiency disorders, are listed as examples.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants were randomly assigned to ozone therapy and placebo groups in a ratio of 1:1 using block randomization with Random Allocation Software (RAS) and block sizes of 4 and 6. By the number of samples, envelopes were prepared, and capsules were deposited within them. 1 to 430 were assigned to each envelope. The envelopes were opened in the order that the participants entered the study, and the type of intervention was determined. A person uninvolved in the sampling process prepared envelopes in the allocation order. In this study, researchers, subjects, and outcome evaluators were all blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of Topical Ozone on The Healing Diabetic Foot Ulcer (Experimental): The topical ozone therapy group received standard wound care with modern dressings every three days for thirty days.
  Interventions: Device: Topical ozone therapy
- Effect of Standart Wound Care on The Healing Diabetic Foot Ulcer (Placebo Comparator): The placebo group received standard wound care with modern dressings thrice weekly for thirty days.
  Interventions: Device: Topical ozone therapy

INTERVENTIONS:
Device: Topical ozone therapy — the topical ozone therapy group received a concentration of 30 mg/L at a frequency of 30 minutes per day for 30 days. Participants received ozone therapy topically every three days for eight treatments.
  Other Names: ozone therapy

SUMMARY:
Despite conflicting and contradictory evidence regarding its efficacy, some wound care centres have advocated and adopted ozone for treating DFU. However, there are gaps in the application of topical ozone therapy. Reported no significant impact on the healing process of DFU, and not all said that topical ozone can enhance the healing process. This study aimed to compare the efficacy of topical ozone therapy in conjunction with standard wound care versus routine wound care alone in treating DFU. The wound, ischemia, and foot infection (WIFI) scale was used to measure wound size, the tissue survival rate at DFU, infection, peripheral microcirculation, glycemic control, Hba1c control, and wound healing.

DETAILED DESCRIPTION:
Diabetic foot ulcer (DFU) is one of the most severe complications that diabetic patients can develop (1). The lifetime incidence of DFUs is estimated to range between 19% and 34%, and between 40% and 65% of diabetic patients experience recurrence within 1 to 5 years after ulcer healing (2). DFUs are prevalent: 6.3% globally and 5.5% in Asia (3). Patients with DFUs have an increased risk of recurrence, infection, necrosis, and ultimately amputation (2-4). The prevalence of diabetic ulcers in Indonesia is around 15%, the amputation rate is 30%, and the mortality rate 1 year after amputation is 14.8% (5). Diabetic foot ulcer patients have a high mortality rate of almost 50% within 5 years with one of the causes being infection (6). The most common reason for hospitalization of people with diabetes is DFU, where 25% are at risk (7) and 20% result in amputations (8). Moreover, according to a meta-analysis, DFU patients in the gangrenous stage have a high risk of amputation (9). DFU treatment costs the healthcare system and the patient's family a lot. DFU control requires specific attention (7). Topical ozone is a cyclic gas composed of three oxygen atoms (10), It can treat various diseases due to its different documented effects, such as its antioxidant and antibacterial properties. Ozone gas treats diseases and wounds, including DFU, in topical ozone therapy (11). Ozone is a gas consisting of three oxygen atoms that decompose swiftly. For instance, it can be used to treat chronic infections primarily caused by pathogens with antibiotic resistance (12).

Study design and participants, in five wound care clinics on Java Island, Indonesia, men and women with diabetic foot ulcer lesions participated in this randomised, triple-blind clinical trial. Inclusion criteria included women and men receiving treatment for diabetic foot ulcers, the WIFI scale, current blood sugar between 120 and 180 mg/dl, Hb1ac between 4.5 and 7%, lesion length greater than 5 cm, and infection. Exclusion criteria in this investigation, such as immunodeficiency disorders, are listed as examples. Sample size, G-Power software was used to calculate the sample size based on the diabetic foot ulcer wound healing variable in the study (11). Taking into account M1 = 39.1, M2 = 33.53, SD1 = 4.4, SD2 = 21.62, = 0.05, and Power = 95%, and taking into account the larger number of samples (n = 210) in each group and 15% attrition, the final sample size for each group was 215, for a total sample size of 430. Sampling, the researcher (first author) enrolled the study with the UHB office of research ethics and awaited a referral letter. Upon entering the room, he introduced himself to the DFU patient, assessed the wound using the WIFI scale, evaluated the inclusion criteria, and explained the purpose and methodologies of the study during wound care. Men and women who were eligible to participate and willing to do so submitted a written consent form. According to their medical records, researchers filled out demographic information. Participants were randomly assigned to ozone therapy and placebo groups in a ratio of 1:1 using block randomization with Random Allocation Software (RAS) and block sizes of 4 and 6. By the number of samples, envelopes were prepared, and capsules were deposited within them. 1 to 430 were assigned to each envelope. The envelopes were opened in the order that the participants entered the study, and the type of intervention was determined. A person uninvolved in the sampling process prepared envelopes in the allocation order. In this study, researchers, subjects, and outcome evaluators were all blinded. Intervention, during wound care, the topical ozone therapy group received a concentration of 30 mg/L at a frequency of 30 minutes per day for 30 days. Participants received ozone therapy topically every three days for eight treatments. The placebo group received standard wound care and education regarding DFU wound care. Both groups received instruction in DFU wound care, personal sanitation, and nutrition. According to the national protocol of the International Working Group on the Diabetic Foot, the same DFU wound care was administered to both groups (13). A document containing a table of the days of the week is provided to the individual, who is instructed to place a mark in the appropriate column each day following consumption. Patients were given a phone number to call if they had any queries or concerns. The degree of wound healing was measured using the Wound, Ischemic, and Edema Infection (WIFI) scale. The enumerator visited each participant at the wound care clinic (data collection and outcome evaluation). Data collection tool, demographic characteristics and the wound, ischemia, foot infection (WIFI) scale were utilised for participant inclusion (14), A summary of adverse events. Age, level of education, employment status, adequate household income, duration of diabetes, course of DFU treatment, number of sutures, blood sugar, Hb1AC, and ankle-brachial index were included as demographic variables (15), and toe ankle brachial (16), dll. Toe ankle brachial Wound, Infection, and Function (WIFI) are graded from 0 to 3. 0: no ulcer, 1: little ulcer, 2: deep ulcer with gangrene limited to toes, 3: extensive ulcer or infection or gangrene. Toe Pressure measures ischemic sites. 0: > 60 mmHg, 1: 40-59, 2: 30-39, 3: <30, while on infection, 0: No infection, 1: Mild (<22cm cellulitis), Moderate (>2cm/purulent), 3: Severe (Systemic response/Sepsis). Data analysis, the collected data were analysed with Jamovi software, and their normality was determined with the Kolmogorov-Smirnov test. Intention-to-treat (ITT) was utilised to analyse the outcomes. In this study, wound healing was regarded as the primary outcome, while infection and ischemia were secondary outcomes. Independent t-test and Multivariate Analysis of Variance (MANOVA) were used to compare the improvements in wound size, brachial toe index, transcutaneous oxygen, and infection between the two groups.

ELIGIBILITY:
Inclusion standarts:

* Patients with diabetic foot ulcers, both male and female, include both sexes.
* Size wound 4-80cm
* Value toe brachial index between 4-7 mmHg
* Value transcutaneous oxygen (TcPO2) levels range 1-45 mmHg
* Infection, area of cellulitis 1-2cm

Exclusion standarts:

* Immunodeficiency conditions
* Concurent ilness
* Size wound >80cm
* Value toe brachial index (TBI) <4 mmHg
* Value crititcal for transcutaneous oxygen (TcPO2) is 0 mmHg
* Systemic infection and sepsis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 430 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the effects of topical ozone therapy and placebo on the healing of diabetic foot ulcers. | Analysis was performed at the Baseline, fifteen days after treatment began, and thirty days after treatment began.
  Comparing the healing of diabetic foot ulcers in the topical ozone therapy group with the control group. The dimensions of a wound can be assessed for wound-healing purposes by employing a photographic apparatus to quantify the length and width of the wound.

SECONDARY OUTCOMES:
Comparison of ischemia to variations in skin oxygen levels by transcutaneous oxygenation (TcPO2) assessment of topical ozone therapy and placebo in diabetic foot ulcers | Analysis was performed at the Baseline, fifteen days after treatment began, and thirty days after treatment began.
  Differences in epidermal oxygenation levels between diabetic foot ulcers treated with topical ozone therapy and those treated with ozone. The utilization of a scale questionnaire (WIFI) for measurement. The measurement of oxygen levels in the skin to assess ischemia can be conducted using transcutaneous oxygen (TcPO2) measurements, employing the PeriFlux 6000 instrument, which provides a measurement scale. In the context of blood pressure, the categorizations are as follows: normal blood pressure is defined as being greater than 45 mmHG, mild blood pressure falls within the range of 40-45 mmHg, moderate blood pressure ranges from 20-39 mmHg, severe blood pressure is within the range of 1-20 mmHg, and critical blood pressure is defined as being at 0 mmHg.
Comparison of improvement in peripheral microcirculation from ischemia in diabetic foot ulcers between topical ozone therapy and a control group using the toe ankle-brachial index (TBI) measurement. | Analysis was performed at the Baseline, fifteen days after treatment began, and thirty days after treatment began.
  Comparing the improvement in peripheral microcirculation of the foot in diabetic foot ulcers treated with topical ozone versus those treated with ozone. The utilization of a scale questionnaire (WIFI) for measurement. Limb ischemia can be assessed by examining the toe brachial index (TBI) using the Vascular Doppler instrument. The TBI is measured on a scale where a value greater than 0.7 mmHg is considered normal, a value between 0.4 and 0.7 mmHg is considered abnormal, and a value below 0.4 mmHg is considered severe. This examination allows for the evaluation of peripheral microcirculation and can help determine the extent of improvement in cases of limb ischemia.
Comparison of topical ozone therapy and placebo groups for diabetic foot ulcer infection | Analysis was performed at the Baseline, fifteen days after treatment began, and thirty days after treatment began
  Comparing the reduction of infection on the surface of diabetic foot ulcers in the groups receiving topical ozone therapy versus those receiving placebo. The utilization of a scale questionnaire (WIFI) for measurement purposes. The reduction in infection was assessed using an ordinal scale that categorized the severity of infection as follows: no infection (0), mild cellulitis measuring 2cm, moderate cellulitis exceeding 2cm, and severe sepsis/systemic infection.

CONTACTS AND LOCATIONS:
Overall Officials: Asmat Burhan, MSN, Study Chair — Universitas of Harapan Bangsa
Locations (1):
- Griya Husada Clinic, Kediri, Indonesia, Indonesia

IPD SHARING:
Plan to Share IPD: No
Only participant data is utilised in this study.

REFERENCES:
- See also: Diabetic foot ulcer is one of the common complications of diabetes disease that is costly and difficult to treat. — https://doi.org/10.1016/j.dsx.2018.11.060
- See also: New classification system for the threatened lower limb, based on the three main factors that have an impact on limb amputation risk: Wound (W), Ischemia (I) and foot Infection ("fI"). — https://doi.org/10.1590/1677-5449.190070
- See also: DFU patients in the gangrenous stage have a high risk of amputation. — https://doi.org/10.1371/journal.pone.0239236
- See also: DFU treatment costs the healthcare system and the patient's family a lot. — http://doi.org/10.1007/s00203-020-01818-x
- See also: Clinical studies have provided evidence on the oxygen-ozone therapy effectiveness in low perfusion syndromes and hyperglycemia, as well as conditions with oxidative stress and inflammation. The oxygen-ozone therapy promotes faster recovery and enhances h — https://doi.org/10.2147/TCRM.S255247
- See also: ozone administration can induce tolerance to oxidative stress and prevent free radical-mediated injury — https://doi.org/10.1186/2045-9912-1-29
- See also: Diabetic foot ulcer patients have a high mortality rate of almost 50% within 5 years with one of the causes being infection — https://doi.org/10.1016/j.amjms.2020.05.012